CLINICAL TRIAL: NCT05990270
Title: The Effect of Education Given to Women on Knowledge, Attitudes and Beliefs on Cervical Cancer
Brief Title: The Effect of Education Given to Women on Cervical Cancer on Knowledge, Attitude and Belief
Acronym: EEWCCKAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Gul OZTAS, PhD, Assist. Prof. Dr, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KahramanmaraşSIUU
Record Dates: First submitted 2023-07-28; First posted 2023-08-14 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2023-07

CONDITIONS: Cancer of Cervix; HPV Infection
Keywords: Cervical cancer,; early diagnosis,; Pap smear,
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; Disease | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): Cervical cancer education will be provided. (The training will be in three sessions, each session will last 20-30 minutes. In the training; ppt presentation for cervical cancer, HPV virus, question and answer method will be used. In addition, female pelvic anatomy, gynecological examination, how the Pap Test is done, and cervical exam on the gynecological examination model. will be explained by showing cancer pathologies ) After the training, the final test data will be obtained by applying the questionnaire again.
  Interventions: Behavioral: education
- control group (No Intervention)

INTERVENTIONS:
Behavioral: education — Cervical cancer education will be provided. (The training will be in three sessions, each session will last 20-30 minutes. In the training; ppt presentation for cervical cancer, HPV virus, question and answer method will be used. In addition, female pelvic anatomy, gynecological examination, how the Pap Test is done, and cervical exam on the gynecological examination model. will be explained by showing cancer pathologies ) After the training, the final test data will be obtained by applying the questionnaire again.
  Arms: EXPERIMENTAL GROUP

SUMMARY:
Aim: The aim of this study is to reveal the effect of education given to women about cervical cancer on knowledge, attitude and belief.

Material and Method: This randomized controlled study was conducted with 130 who had a public hospital located in Southeast Turkey (51 experimental, 51 control).

DETAILED DESCRIPTION:
Aim: The aim of this study is to reveal the effect of education given to women about cervical cancer on knowledge, attitude and belief.

Material and Method: This randomized controlled study was conducted with 130 who had a public hospital located in Southeast Turkey (51 experimental, 51 control).

In the first stage, the researcher participants were informed about the purpose of the researcher and the questionnaire, and their consent was obtained for participation in the study.

In the second stage, pre-test data will be obtained with the face-to-face interview method of the research data and a questionnaire form. Cervical cancer education will be provided. (The training is in three sessions, each session will last 20-30 minutes. In the training; Cervical cancer, ppt presentation on HPV virus, question-answer method, female pelvic anatomy on the gynecological examination model, gynecological examination, how the Pap Test is done, and cervical cancer pathologies. will be explained )) After the training, the post-test data will be obtained by applying the questionnaire again.

ELIGIBILITY:
Inclusion Criteria:

* least literate, no communication problem women who agreed to participate in the study

Exclusion Criteria:

* literate are women who do not have communication problems (hearing impairment, visual impairment)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
First Measurement: Human Papilloma Virus (HPV) Knowledge Scale | Measurement at the second encounter (1 WEEK AFTER TRAINING) for each group.
  ASSESSMENT OF WOMEN'S AWARENESS ON HPV
Second Measurement:Cervical Cancer and Pap-Smear Test Health Belief Model Scale | Measurement at the second encounter (1 WEEK AFTER TRAINING) for each group.
  ASSESSMENT OF HEALTH BELIEFS

CONTACTS AND LOCATIONS:
Overall Officials: HATİCE GÜL ÖZTAŞ, Study Director — KahramanmaraşISU
Locations (1):
- Kahramanmaraş ISU, Kahramanmaraş, K.Maraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gul Oztas H, Isik K. The Effect of Cervical Cancer Education Given to Women in Turkey on Knowledge, Attitudes, and Health Beliefs: A Randomized Controlled Study. Public Health Nurs. 2025 Jan-Feb;42(1):363-373. doi: 10.1111/phn.13456. Epub 2024 Oct 17. PMID 39420668